CLINICAL TRIAL: NCT03727334
Title: Offsetting Hippocampal Degeneration in Moderate to Severe TBI
Brief Title: Offsetting Hippocampal Degeneration in m-sTBI
Acronym: m-sTBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, William Panenka, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H17-03544
Record Dates: First submitted 2018-10-03; First posted 2018-11-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Traumatic Brain Injury; Degeneration; Memory; Loss, Mild, Following Organic Brain Damage
MeSH Terms: conditions — Brain Injuries, Traumatic; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: This is a randomized two-armed study, comprised of a treatment arm and a control arm. Given the small numbers and the potentially slow rate of recruitment, the investigators will employ simple rather than block randomization. To minimize selection bias, allocation to group will be concealed (i.e., with assignment unpredictable and unchangeable) using software that randomizes each patient upon confirmation of eligibility. Patients will not be blind to group assignment, but the psychometrist completing behavioural outcomes will be kept blind to group assignment.
Who Masked: Outcomes Assessor
Masking Description: The psychometrist will be blind to the arm the participant is assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): For the treatment arm, the participants will complete the intervention protocol following the first in-person study visit 7 months post-injury. The intervention involves 16 weeks of online, in-home spatial navigation training. During the 16 weeks, the participant will complete exercises for 1 hour/day, 5 days a week.
  Interventions: Behavioral: Online Spatial Navigation Training
- Control (No Intervention): The control arm participants will receive their typical standard of care; they will not complete the intervention but will complete all of the in-person visits at the same post-injury time-points as the treatment group.

INTERVENTIONS:
Behavioral: Online Spatial Navigation Training — Participants complete training tasks that test their spatial navigational abilities, cognitive map formation, and pattern separation. These training tasks involve map drawing, vector mapping, proximity judgments, and navigating with blocked routes.
  Arms: Treatment

SUMMARY:
The goal of this study is to establish the feasibility of an intervention designed to improve memory in patients who have experienced a moderate or severe traumatic brain injury (m-sTBI) and to examine its effect on brain structures.

DETAILED DESCRIPTION:
The purpose of this study is to establish the feasibility of a novel intervention, and explore biomarker predictors of neurodegeneration and response to the proposed intervention. This 16 week intervention utilises allocentric spatial navigation tasks to improve memory and counteract hippocampal neurodegeneration. This intervention will be administered in combination with neuropsychological assessments, MR imaging, and the analysis of genomic variants at two time points; 7 months post-TBI and 12 months post-TBI.

ELIGIBILITY:
Inclusion Criteria:

* An acute care diagnosis of TBI as determined by a medical professional, indicated by:

  * Post-traumatic amnesia duration of 24 hours or more, and/or lowest Glasgow Coma Scale score of < 13
  * Positive clinical CT or MRI scan
* Aged 18 to 65
* Fluent in English
* Have the competency for fully informed consent by 6 months post-injury
* Have basic computer skills
* Have functional use of one upper extremity
* Have access to the internet

Exclusion Criteria:

* A neurological disorder other than TBI (e.g., stroke, dementia, tumor, neurodevelopmental disorder) impairing baseline awareness, cognition, or validity of follow-up and outcome assessment.
* A systemic condition (e.g., lupus, diabetes, rheumatoid arthritis).
* Any contraindications to magnetic resonance imaging (MRI)
* You are experiencing language impairments (i.e., aphasia) from your injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Online Spatial Navigation Intervention Test Scores: Change in Spatial Learning Ability | Time-point 1: 7 months post-injury and Time-point 2: 12 months post-injury
  Participants complete online spatial navigation training 5 days per week for 16 weeks. Improvement in spatial learning ability will be assessed based on the accuracy of answers to questions regarding the reproduction of spatial elements, the direction and proximity of certain landmarks, and describing the most efficient route from point A to point B. Improvement will be assessed at the end of each week and at the end of the intervention. The raw scores range from 0-15, with higher scores indicating better spatial learning ability.
Online Spatial Navigation Intervention Test Scores: Change in Cognitive Map Formation | Time-point 1: 7 months post-injury and Time-point 2: 12 months post-injury
  Participants complete online spatial navigation training 5 days per week for 16 weeks. Improvement in cognitive map formation will be assessed based on the number of trails required by the participant to learn landmark placements and based on the accuracy of the participant's navigation to a specific destination. The raw scores range from 1-21 and 0-10, respectively. A decrease in the number of trials required by the participant and an increase in navigation accuracy both correspond to an improvement in cognitive map formation.
Online Spatial Navigation Intervention Test Scores: Change in Pattern Separation | Time-point 1: 7 months post-injury and Time-point 2: 12 months post-injury
  Measurement of pattern separation abilities are assessed in a task requiring the participant to differentiate memories in order to prevent interference from overlapping details. The following three variables are taken into account: i) percent correct ii) the discriminating value and iii) bias metric. Percent correct and bias metric are given as a percentage values (e.g., 80.63%) and the discriminating variable is given as a raw rate (e.g., 0.67). An improvement in pattern separation abilities are determined by an increase in percent correct and discrimination values from pre- to post-intervention. An increase in bias metric from pre- to post-intervention reflects an increased tendency for pattern separation.
Online Spatial Navigation Intervention Test Scores: Change in Pattern Completion | Time-point 1: 7 months post-injury and Time-point 2: 12 months post-injury
  Measurement of pattern completion abilities are assessed in a task designed to probe pattern completion by presenting partial retrieval cues at different levels of degradation. The following variables are taken into account: i) accuracy for learned stimuli given as a percentage value (i.e., correctly selecting the name of the scene) ii) accuracy for new stimuli given as a percentage value (i.e., correctly indicating the stimuli is novel) and iii) bias measure. The bias measure is obtained by subtracting the learned stimuli accuracy score from the new stimuli accuracy score. An increase for both accuracy measures from pre- to post-intervention corresponds to improvement on recognition memory. An increase in bias measure reflects an increased tendency for pattern separation.

SECONDARY OUTCOMES:
Neuronal injury biomarker predictors in serum and plasma samples | Time-point 1: 7 months post-injury and Time-point 2: 12 months post-injury
  The investigators will be analysing biomarkers in serum and plasma samples in relation to traumatic brain injuries. This will allow the investigators to generate hypotheses concerning the relationship between blood biomarkers and neuronal injury. Serum neurofilament light chains (NF-L), total tau, amyloid β-40 and amyloid β-42 will be assayed using Quanterix reagents on the Simoa HD-1 platform.
Gliosis and inflammation biomarker predictors in serum samples | Time-point 1: 7 months post-injury and Time-point 2: 12 months post-injury
  The investigators will be analysing biomarkers in serum samples in relation to gliosis and inflammation. This will allow the investigators to generate hypotheses concerning the relationship between blood biomarkers and neuroimmune response. Serum monocyte chemoattractant protein-1 (MCP-1) will be assayed using MesoScale Discovery reagents on the Sector S600 platform and glial fibrillary acidic protein (GFAP) will be assayed using Quanterix reagents on the Simoa HD-1 platform.

CONTACTS AND LOCATIONS:
Overall Officials: William Panenka, MD, Principal Investigator — University of British Columbia; Robin Green, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Vancouver General Hopsital, Vancouver, British Columbia
  - GF Strong Rehabilitation Centre, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No